CLINICAL TRIAL: NCT04978649
Title: Intervention for High-normal Blood Pressure in Adults With Type 2 Diabetes-----renal Substudy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Cooperation plan has been changed
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, XueQing Yu, Dean, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GDPH-IPAD-CKD
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2; Blood Pressure
Keywords: prehypertension; renal disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prehypertension; Kidney Diseases | interventions — allisartan isoproxil; Amlodipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensive treatment group (Active Comparator): Real antihypertensive agents will be provided for this arm, to decrease systolic BP to lower than 120 mm Hg. In this group, the following study medications will be used: tablets with Allisartan Isoproxil 240 mg (first-line medication); tablets with Amlodipine 5 mg (second-line medication). Treatment will be started with Allisartan 240 mg. If necessary to reach the BP goal, Amlodipine (first 5 mg or then 10 mg daily) will be given in addition. If intolerable side effects occur, first-line medication may be replaced by second-line medication.
  Interventions: Drug: Allisartan Isoproxil; Drug: Amlodipine
- standard treatment group (Placebo Comparator): In this arm participants are followed up and no medications be used until BP becomes ≥ 140 mm Hg systolic and/or 90 mm Hg diastolic. Medications are determined by investigators in lines with recommendations by current Chinese guidelines to decrease BP to lower than 140 mm Hg systolic and to lower than 90 mm Hg diastolic.
  Interventions: Drug: Allisartan Isoproxil; Drug: Amlodipine

INTERVENTIONS:
Drug: Allisartan Isoproxil — Allisartan Isoproxil 240mg daily will be used to lower BP to below 120 mm Hg systolic.
  Other Names: Xinlitan
Drug: Amlodipine — Amlodipine 5mg daily will be added to Allisartan Isoproxil and afterwards increased to 10mg daily, if necessary to reach the blood pressure goal (below 120 mm Hg systolic).
  Other Names: Qiaohean

SUMMARY:
Lowering of blood pressure (BP) in high-risk hypertensive individuals reduces major adverse cardiovascular (CV) and renal events. Diabetic patients with hypertension benefit from BP lowering treatment. The present trial, IPAD-CKD in brief, is a randomized, open-label, parallel-designed, multicenter study involving nearly 5322 patients to be recruited over three years and to be followed up for a median of four years and a half. IPAD-CKD tests the hypothesis that antihypertensive medications in adults with type 2 diabetes, whose seated BP 120-139 mm Hg systolic and below 90 mm Hg diastolic, results in 20% difference in the incidence of major renal events. During follow-up for participants in the intensive group, the sitting systolic pressure should be decreased to below 120 mm Hg, by titration and combination of the double-blind study medications of an angiotensin type-1 receptor blocker Allisartan (240 mg/day), a dihydropyridine calcium-channel blocker (amlodipine 5-10 mg/day), and/or other medications if necessary. For those in the standard group, the sitting systolic pressure should be monitored and controlled below 140 mm Hg.

DETAILED DESCRIPTION:
The IPAD-CKD trial is a randomized, open-label, parallel-designed, multicenter study. 5322 patients will be recruited over three years with a median follow up of 4.5 years. IPAD tests the hypothesis that intensive antihypertensive medical therapy in adult patients with type 2 diabetes, whose seated BP ranges from 120 to 139 mm Hg systolic and < 90 mm Hg diastolic, results in 20% reduction in the incidence of major renal events (the primary endpoint), a composite of renal failure and proteinuria progression. Secondary endpoints of this study include: renal failure ; proteinuria progression; proteinuria reversion; end stage renal disease; cardiovascular-cause mortality; MI; hospitalization for HF; stroke;hospitalization for unstable angina; all-cause mortality;development of diabetic retinopathy that needs interventional operation; peripheral arterial diseases; new on-set atrial fibrillation or flutter; cancer.

Inclusion criteria for the study include T2DM patients aged between 45 and 79 years within the aforementioned BP ranges. For participants in the intensive group, the sitting systolic BP should decrease to < 120 mm Hg, using titration and combination of study medications consisting of an angiotensin type-1 receptor blocker Allisartan (240 mg/day) and a dihydropyridine calcium-channel blocker (amlodipine 5-10 mg/day), and/or other medications if necessary.For those in the standard group, the sitting systolic pressure should be monitored and controlled below 140 mm Hg. Across the whole study, 310 primary endpoints are expected to occur. Interim analyses will be carried out on an intention-to-treat basis at the accumulation of 107 and 214 primary endpoints respectively. At the completion of the trial, both an intention-to-treat and a per-protocol analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* irrespective of sex;
* aged between 45 and 79 years;
* with office-measured seated BP 120-139 mm Hg systolic and below 90 mm Hg diastolic;
* diagnosed of type 2 diabetes mellitus (T2DM), currently on diabetic therapy; a glycosylated hemoglobin (HbA1c) ≤ 8.5%;
* informed consent provided and long-term follow-up possible

Exclusion Criteria:

* administration of any antihypertensive medications within 1 month;
* a history of hypoglycemic coma / seizure;
* confirmed diagnosis of type 1 diabetes mellitus;
* alanine-aminotransferase (ALT) or aspartate-aminotransferase (AST) over three times the upper limit of normal;
* estimated glomerular filtration rate < 45 ml/min/1.73m2;
* a history of congestive heart failure with left ventricular ejection fraction < 40%, requiring treatment with renin-angiotensin system (RAS) blockers; coronary artery disease requiring RAS blockers for secondary prevention;
* acute on-set of stroke within 6 months prior to randomization;
* a ratio of urinary albumin (in mg/L) to urinary creatinine (in g/L) (ACR) ≥ 300 mg/g;
* a history of primary or secondary renal diesease requiring a therapy using glucocorticoid or immunity inhibitor;
* a history of polycystic kidney;
* known contraindications for the active study medications;
* a history of psychological or mental disorder;
* pregnancy or currently planning to have babies or lactation;
* severe diseases such as severe valvular heart diseases;
* an expected residual life span less than 3 years;
* a malignancy that clinical investigators consider as unsuitable to participate;
* currently participating in another clinical trial.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Major Renal Events | From date of randomization until the date of first documented incidence of the major renal events prespecified, whichever comes first, assessed up to 60 months
  The major renal events defined in the study include a composite of renal failure (defined as dialysis, transplantation, or a sustained estimated GFR of <15 ml per minute per 1.73 m 2), or serum creatinine level >3.3 mg/dl, or a doubling of the serum creatinine level）and proteinuria progression（defined as:uACR ≥30 mg/gCr if baseline uACR< 30 mg/gCr; uACR ≥300 mg/gCr if baseline uACR is between 30 to 300 mg/gCr.
  ）

SECONDARY OUTCOMES:
renal failure | From date of randomization until the date of first documented incidence of the major renal events prespecified, whichever comes first, assessed up to 60 months
  dialysis, transplantation, or a sustained estimated GFR of <15 ml per minute per 1.73 m 2), or serum creatinine level >3.3 mg/dl, or a doubling of the serum creatinine level
proteinuria progression | From date of randomization until the date of first documented incidence of the major renal events prespecified, whichever comes first, assessed up to 60 months
  uACR ≥30 mg/gCr if baseline uACR< 30 mg/gCr; uACR ≥300 mg/gCr if baseline uACR is between 30 to 300 mg/gCr.
proteinuria reversion | From date of randomization until the date of first documented incidence of the major renal events prespecified, whichever comes first, assessed up to 60 months
  uACR <30mg/gCr if baseline uACR is between 30 to 300 mg/gCr.
cardiovascular-cause mortality | From date of randomization until the date of first documented incidence of the major renal events prespecified, whichever comes first, assessed up to 60 months
  Cardiovascular death include death caused by stroke, MI, HF, sudden death or any other death attributed to cardiovascular diseases. Sudden death (ICD-Code I46.1, R96) encompasses any death of unknown origin occurring instantly or within an estimated 24 hours after the onset of acute symptoms as well as unattended death for which no likely cause can be established by autopsy or recent medical history.
Acute Myocardial Infarction | From date of randomization until the date of first documented incidence of the major renal events prespecified, whichever comes first, assessed up to 60 months
  Acute myocardial infarction (MI) is defined when any one of the following criteria occurs. (1) Detection of a rise and/or fall of cardiac biomarker values, with at least one value above the 99th percentile upper reference limit and with at least one of the following manifestations: symptoms of ischaemia that should have lasted for at least 30 minutes and should not have been responsive to sublingual administration of nitrates; new or presumed new significant ST-segment-T wave changes or new left bundle branch block (LBBB); development of pathological Q waves in the ECG; imaging evidence of new loss of viable myocardium or new regional wall motion abnormality. (2) Identification of an intracoronary thrombus by angiography or autopsy. (3) Cardiac death with symptoms suggestive of myocardial ischaemia and presumed new ischaemic ECG changes or new LBBB, but death occurred before cardiac biomarkers were obtained, or before cardiac biomarker values would be increased.
Hospitalization of Congestive Heart Failure | From date of randomization until the date of first documented incidence of the major renal events prespecified, whichever comes first, assessed up to 60 months
  Congestive heart failure (HF) requires the presence of three conditions, namely symptoms, such as dyspnea, clinical signs, such as ankle edema or crepitations, and the necessity to initiate treatment with open-label diuretics, vasodilators or antihypertensive drugs. HF cases may also be adjudicated as chronic stable HF but this is not considered an outcome of the present study.
Hospitalization of Unstable Angina | From date of randomization until the date of first documented incidence of the major renal events prespecified, whichever comes first, assessed up to 60 months
  Unstable angina is defined as new onset or worsening angina pectoris requiring hospitalization with angiographically documented coronary atherosclerosis or transient electrocardiographic changes of the ST-segment or T-wave without evidence for myocardial necrosis. This diagnosis excludes patients with angina pectoris admitted to the hospital only for investigation.
All-cause Mortality | Time Frame: From date of randomization until the date of death from any causes, assessed up to 60 months.
  All-cause mortality refers to death from any causes.
Diabetic Retinopathy Requiring Interventional Operation or Surgery | Time Frame: From date of randomization until the date of death from any causes, assessed up to 60 months.
  Diabetic retinopathy requiring interventional operation or surgery is defined as the confirmed diagnosis of diabetic retinopathy, indicated for interventional operation or surgery, which is documented by ophthalmologists.
Peripheral Arterial Diseases Requiring Revascularization | Time Frame: From date of randomization until the date of death from any causes, assessed up to 60 months.
  Peripheral arterial diseases requiring revascularization are defined as the confirmed diagnosis of any one of the peripheral arterial diseases indicated for revascularization.
New Atrial Fibrillation or Flutter | Time Frame: From date of randomization until the date of death from any causes, assessed up to 60 months.
  Atrial fibrillation or flutter is confirmed and documented with electrocardiogram indicating the occurence of atrial fibrillation or flutter. New development of atrial fibrillation or flutter is defined only if a participant at baseline has no history of and his or her electrocardiogram shows no signs of atrial fibrillation or flutter.
Cancer | Time Frame: From date of randomization until the date of death from any causes, assessed up to 60 months.
  Cancer defined in the present study is recorded only when there is pathologically confirmed evidence.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, Doctor, Study Chair — Guangdong Provincial People's Hospital